CLINICAL TRIAL: NCT07297654
Title: First-Line Lenvatinib in Child-Pugh B Patients With HCC Unsuitable for Curative Treatment: A Phase 2 FINELAND Trial
Brief Title: First-Line Lenvatinib in Child-Pugh B Patients With HCC Unsuitable for Curative Treatment
Acronym: FINELAND
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Center, Korea (Other Government)
Collaborators: Asan Medical Center (Other); Seoul National University Hospital (Other); Seoul National University Bundang Hospital (Other); Samsung Medical Center (Other); Hanyang University Guri Hospital (Other)
Responsible Party: Principal Investigator, Bo Hyun Kim, Principal Investigator, National Cancer Center, Korea
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC2025-0327
Record Dates: First submitted 2025-12-09; First posted 2025-12-22 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Advanced Hepatocellular Carcinoma
Keywords: Lenvatinib; child Pugh B
MeSH Terms: interventions — lenvatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lenvatinib (Experimental): Lenvatinib will be administered orally once daily at a dose of 8 mg, at the same time each day, with or without food.
  Treatment must begin within 3 days after screening and will continue until disease progression, unacceptable toxicity, withdrawal of consent, or study termination, whichever occurs first.
  Interventions: Drug: Lenvatinib

INTERVENTIONS:
Drug: Lenvatinib — Lenvatinib will be administered orally at a dose of 8 mg once daily at the same time each day, with or without food (regardless of body weight). For participants with a baseline body weight ≥60 kg who tolerate lenvatinib at 8 mg once daily (i.e., experiencing only Grade 1 or lower adverse events) and have maintained this dose for at least 2 weeks, the daily dose of lenvatinib may be increased to 12 mg.

SUMMARY:
This study aims to evaluate the efficacy and safety of lenvatinib as first-line therapy in patients with Child-Pugh class B HCC who are unsuitable for curative treatment.

DETAILED DESCRIPTION:
<Treatment Phase> All participants will receive lenvatinib treatment after signing informed consent. Lenvatinib will be administered orally once daily at a dose of 8 mg, at the same time each day, with or without food.

Treatment must begin within 3 days after screening and will continue until disease progression, unacceptable toxicity, withdrawal of consent, or study termination, whichever occurs first.

<Follow-up Phase> After the treatment phase, participants will be followed every 12 weeks (±7 days) after the last dose for survival status and use of subsequent anticancer therapies. Survival follow-up will be conducted for at least 12 months after enrollment of the last participant.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Age ≥ 19 years at the time of signing informed consent
3. Histological or clinical diagnosis of HCC according to the Korean Liver Cancer Association-National Cancer Center guidelines
4. HCC not amenable to curative treatment (e.g., surgical resection, local therapy, liver transplantation)
5. At least one measurable target lesion according to RECIST v1.1

   - Participants who previously received local treatment (e.g., radiofrequency ablation, microwave ablation, transarterial chemoembolization, transarterial radioembolization, transarterial embolization, or radiotherapy) are eligible if (a) target lesions have not been treated by prior local therapy, or (b) lesions within the field of local therapy have subsequently progressed according to RECIST v1.1.
6. Child-Pugh class B7-B8
7. ECOG performance status (PS) 0-2
8. Adequate hematologic and end-organ function defined by the following laboratory tests obtained within 14 days prior to screening:

   * Hemoglobin ≥ 8.0g/dL
   * Absolute neutrophil count (ANC) ≥ 1,000/mm3
   * Platelet count ≥ 50,000/μL
   * Total bilirubin < 3.5 mg/dL
   * Serum albumin ≥ 2.5 g/dL
   * ALT and AST ≤ 7 x upper limit of normal (ULN)
   * Prothrombin time (INR ≤ 1.8 × ULN)
   * Serum creatinine ≤ 2.0 × ULN or calculated creatinine clearance ≥ 40 mL/min (Cockcroft-Gault equation)
9. Documented virological status for hepatitis B virus (HBV) and hepatitis C virus (HCV) by screening tests.

   - Participants with HBV or HCV infection must receive antiviral therapy in accordance with institutional guidelines.
10. Women of childbearing potential must agree to remain abstinent or use effective contraception (failure rate < 1% per year) from signing informed consent through at least 6 months after the last study drug administration.

Men must agree to remain abstinent or use effective contraception (failure rate < 1% per year) during the same period and refrain from sperm donation.

Exclusion Criteria:

1. Fibrolamellar carcinoma or sarcomatoid carcinoma
2. Prior systemic therapy for HCC
3. Local therapy for HCC (including radiofrequency ablation, microwave ablation, cryoablation, transarterial chemoembolization, radioembolization, or radiotherapy) within 28 days prior to initiation of study treatment, or unresolved complications from such procedures

   - Palliative radiotherapy to bone lesions is permitted with a 7-day washout
4. History of allogeneic stem cell or solid organ transplantation
5. Active brain metastases or leptomeningeal disease
6. History of another malignancy within 2 years prior to screening, except for cancers with negligible risk of metastasis or death (e.g., >90% 5-year survival)
7. Serious uncontrolled medical comorbidities within 3 months prior to study treatment, including severe cardiovascular disease (NYHA class ≥ II heart disease, myocardial infarction, or cerebrovascular accident), unstable arrhythmia, or unstable angina, or any condition judged by the investigator to increase participant risk
8. Pregnant or breastfeeding women, or men and women of reproductive potential unwilling to use effective contraception from screening through 6 months after the last study drug administration
9. Any condition judged by the investigator to interfere with compliance with study procedures, restrictions, or requirements

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Twelve months after the last subject is enrolled or the time at which the 41 events required to verify the assumptions used in the sample size calculation have occurred
  Progression-free survival (PFS) is defined as the time from the date of treatment initiation to the date of first documented progressive disease (PD) according to RECIST v1.1, as assessed by the investigator, or death from any cause.

SECONDARY OUTCOMES:
Overall survival (OS) | Twelve months after the last subject is enrolled or the time at which the 41 events required to verify the assumptions used in the sample size calculation have occurred
  Overall survival (OS) is defined as the time from the date of treatment initiation to death from any cause.
Time to progression (TTP) | Twelve months after the last subject is enrolled or the time at which the 41 events required to verify the assumptions used in the sample size calculation have occurred.
  Time to progression (TTP) is defined as the time from the date of treatment initiation to the date of first documented progressive disease (PD) according to RECIST v1.1, as assessed by the investigator.
Objective response rate (ORR) | Twelve months after the last subject is enrolled or the time at which the 41 events required to verify the assumptions used in the sample size calculation have occurred.
  Objective response rate (ORR) is defined as the proportion of participants whose best overall response is complete response (CR) or partial response (PR), as assessed by the investigator according to RECIST v1.1.
Disease control rate (DCR) | Twelve months after the last subject is enrolled or the time at which the 41 events required to verify the assumptions used in the sample size calculation have occurred.
  Disease control rate (DCR) is defined as the proportion of participants whose best overall response is complete CR, PR, or stable disease (SD), as assessed by the investigator according to RECIST v1.1.
The incidence of AEs | Twelve months after the last subject is enrolled or the time at which the 41 events required to verify the assumptions used in the sample size calculation have occurred.
  The incidence of AEs is defined as the number of all AEs occurring in participants from the first dose of the investigational product until the last follow-up visit, as well as the proportion of participants who experience them. The severity of AEs will be graded on a scale of Grade 1-5 according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Bo Hyun Kim Kim, MD, Principal Investigator — National Cancer Center

IPD SHARING:
Plan to Share IPD: Undecided